CLINICAL TRIAL: NCT06521515
Title: The Impact of Lung Ultrasound Morphology Patterns on Treatment Response and Weaning Outcomes in High-Risk Mechanically Ventilated Patients
Brief Title: Lung Ultrasound Morphology Patterns Predict Weaning Outcomes
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LUMP-WO
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Retrospective
Keywords: weaning; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TLP group: Patients were grouped into TLP if they exhibited a tissue-like pattern in any region
  Interventions: Diagnostic Test: Lung Ultrasound Morphology Patterns
- DBP group: Patients were grouped into DBP if they displayed diffuse B-lines and shred signs in most regions.
  Interventions: Diagnostic Test: Lung Ultrasound Morphology Patterns

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound Morphology Patterns — Two blinded investigators conducted daily lung ultrasound examinations. Each lung was scanned in six regions, categorizing ultrasound findings into four aeration patterns: normal (N-score 0), moderate (B1-lines score 1), severe (B2-lines score 2), and consolidation (C-score 3). The global LUS score ranged from 0 to 36. Patients were grouped into TLP if they exhibited a tissue-like pattern in any region or DBP if they displayed diffuse B-lines and shred signs in most regions. Localized TLPs indicated concentrated areas of non-aeration.

SUMMARY:
This prospective observational study aims to investigate the impact of lung ultrasound morphology patterns on treatment response and weaning outcomes in high-risk mechanically ventilated patients. The study will be conducted in the intensive care unit (ICU) and will include patients who have been on mechanical ventilation for over 24 hours, are at high risk for reintubation due to age (>65 years) or underlying conditions (chronic heart or lung disease), and have a Lung Ultrasound Score (LUS) >13.

Patients will be stratified into two groups based on their lung ultrasound patterns: localized tissue-like patterns (TLP) and diffuse B-lines (DBP). Daily lung ultrasound examinations will be performed, and patients will receive targeted clinical interventions based on their ultrasound findings, such as lung recruitment maneuvers, positive end-expiratory pressure (PEEP) ventilation, prone positioning, pleural effusion drainage, antibiotics for pneumonia, and strategies for achieving negative fluid balance.

The primary outcome will be the change in Lung Recruitment Score (LRS) between the TLP and DBP groups, which assesses lung recruitment efficiency. Secondary outcomes will include the rate of weaning failure, duration of mechanical ventilation, ICU mortality, total ICU stay duration, and PaO2/FiO2 ratio before and after the spontaneous breathing trial (SBT).

This study aims to provide insights into the utility of lung ultrasound morphology patterns in guiding clinical interventions and predicting weaning outcomes in high-risk mechanically ventilated patients, potentially leading to improved patient care and outcomes in the ICU setting.

DETAILED DESCRIPTION:
This prospective observational study, titled "Lung Ultrasound Morphology Patterns Predict Weaning Outcomes (LUMP-WO)," aims to investigate the impact of lung ultrasound morphology patterns on treatment response and weaning outcomes in high-risk mechanically ventilated patients. The study will be conducted in the intensive care unit (ICU) of a tertiary care hospital.

Inclusion criteria for the study are: (1) mechanical ventilation for over 24 hours before the first spontaneous breathing trial, (2) high risk for reintubation due to age (>65 years) or underlying conditions (chronic heart disease or chronic lung disease), and (3) complete ultrasound data and initial LUS score >13. Exclusion criteria include: (1) age under 18 years, pregnancy, mechanical ventilation duration less than 24 hours, or diaphragmatic dysfunction; (2) low risk of extubation failure; (3) peripheral neuromuscular disorders; or (4) do-not-reintubate order at the first spontaneous breathing trial.

Patients will undergo daily lung ultrasound examinations performed by blinded investigators. Each lung will be scanned in six regions, and ultrasound findings will be categorized into four aeration patterns: normal (N-score 0), moderate (B1-lines score 1), severe (B2-lines score 2), and consolidation (C-score 3). The global LUS score will range from 0 to 36. Patients will be grouped into TLP if they exhibit a tissue-like pattern in any region or DBP if they display diffuse B-lines and shred signs in most regions.

Patients will receive standard medical care and targeted interventions based on their lung ultrasound findings. Lung recruitment maneuvers, PEEP ventilation, prone positioning, pleural effusion drainage, antibiotics for pneumonia, and strategies for achieving negative fluid balance will be utilized as appropriate. Weaning criteria will be assessed daily, and the Spontaneous Breathing Test (SBT) will be conducted using a T-tube or mechanical ventilation with low PEEP and pressure support.

The primary outcome will be the change in Lung Recruitment Score (LRS) between the TLP and DBP groups. Secondary outcomes will include the rate of weaning failure, duration of mechanical ventilation, ICU mortality, total ICU stay duration, and PaO2/FiO2 ratio before and after the SBT.

Data will be analyzed using appropriate statistical tests, and univariate and multivariate regression analyses will be utilized to identify risk factors associated with weaning outcomes.

This study aims to provide valuable insights into the utility of lung ultrasound morphology patterns in guiding clinical interventions and predicting weaning outcomes in high-risk mechanically ventilated patients. The findings may contribute to the development of personalized management strategies and improved patient outcomes in the ICU setting. The study's results may also help in the early identification of patients at risk of weaning failure, allowing for timely interventions and resource allocation.

ELIGIBILITY:
Inclusion criteria:(1) age ≥18 years, (2) on mechanical ventilation >24 hours before the first spontaneous breathing trial, (3) high risk for reintubation due to age (>65 years) or chronic heart or lung disease, and (4) complete ultrasound data and initial LUS >13.

Exclusion criteria:(1) age under 18 years, pregnancy, mechanical ventilation duration less than 24 hours, or diaphragmatic dysfunction; (2) low risk of extubation failure; (3) peripheral neuromuscular disorders; or (4) do-not-reintubate order at the first spontaneous breathing trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be retrospective. Based on lung ultrasound morphology patterns, patients will be stratified into localized tissue-like patterns (TLP) and diffuse B-lines (DBP) groups. The study will enroll a diverse population to ensure generalizability and comprehensively analyze the relationship between lung ultrasound morphology patterns, treatment response, and weaning outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
LRS | through study completion，up to 28 days
  The primary endpoint of the study was the change in Lung Recruitment Score (LRS) between the TLP and DBP groups. LRS assesses lung recruitment efficiency, assigning positive scores for reaeration and negative scores for loss of aeration (

SECONDARY OUTCOMES:
weaning failure rates | through study completion,up to 28 days
  defined as inability to successfully complete a spontaneous breathing trial, need for mechanical ventilation reintroduction within 48 hours post-weaning, or mortality related to weaning.
duration of mechanical ventilation | through study completion,up to 28 days
  the total number of days or hours a patient receives invasive mechanical ventilation support
ICU mortality | through study completion,up to 28 days
  the proportion of patients who die during their stay in the intensive care unit (ICU).
total ICU stay duration | through study completion,up to 28 days
  the number of days a patient remains in the ICU from admission to discharge, transfer to another unit, or death.
PaO2/FiO2 ratio before and after the spontaneous breathing trial (SBT) | through study completion,up to 28 days
  The PaO2/FiO2 ratio will be calculated by dividing the partial pressure of arterial oxygen (PaO2) by the fraction of inspired oxygen (FiO2). Measurements will be taken at two time points: (1) immediately before the start of the SBT and (2) at the end of the SBT or at the time of SBT failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, Ph.D, Study Chair — Fudan University
Locations (1):
- Hongyu He, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) sharing plan for this study will involve making specific datasets available to other researchers upon request and after the publication of the primary study results. The IPD to be shared will include de-identified data on patient demographics, clinical characteristics, lung ultrasound findings, treatment interventions, and outcomes, such as the duration of mechanical ventilation, ICU mortality, total ICU stay duration, and PaO2/FiO2 ratio before and after the spontaneous breathing trial (SBT).
Supporting Information: Study Protocol
Time Frame: After the publication of the primary study results, the IPD will be available for request by other researchers for a period of 6 to 36 months.
Access Criteria: Researchers interested in obtaining the IPD must submit a written application, detailing the research purpose, proposed analysis plan, and data usage and protection plan. All applications will be reviewed by the research team to ensure that the proposed research is consistent with the informed consent provided by the original study participants and complies with relevant ethical and regulatory requirements. Access to the IPD may require the execution of a data use agreement to stipulate the terms of data usage, storage, sharing, etc.

REFERENCES:
- [Result] Bello G, Blanco P. Lung Ultrasonography for Assessing Lung Aeration in Acute Respiratory Distress Syndrome: A Narrative Review. J Ultrasound Med. 2019 Jan;38(1):27-37. doi: 10.1002/jum.14671. Epub 2018 May 6. PMID 29732586
- [Result] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Result] Mayo P, Volpicelli G, Lerolle N, Schreiber A, Doelken P, Vieillard-Baron A. Ultrasonography evaluation during the weaning process: the heart, the diaphragm, the pleura and the lung. Intensive Care Med. 2016 Jul;42(7):1107-17. doi: 10.1007/s00134-016-4245-3. Epub 2016 Mar 7. PMID 26951426